CLINICAL TRIAL: NCT05868928
Title: Imaging Risks for Recurrence After Stereotactic Radiosurgery in Brain Metastasis (IRRAS-BM)
Brief Title: Imaging Features for the Risks for Recurrence After Stereotactic Radiosurgery in Brain Metastasis
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Professor, Asan Medical Center
Other Study IDs: AsanMCHSKim_07
Record Dates: First submitted 2023-04-16; First posted 2023-05-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Brain Metastases; Radiosurgery
Keywords: Imaging; Habitat; Recurrence; Prediction; Radiation necrosis
MeSH Terms: conditions — Brain Neoplasms; Recurrence | interventions — Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain metastases patients who received stereotactic radiosurgery: Patients with brain metastases who received stereotactic radiosurgery
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Diffusion-weighted MRI; Diagnostic Test: Arterial spin labeling (ASL); Diagnostic Test: Dynamic susceptibility contrast-MRI (DSC-MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — Pre-and post-contrast enhanced T1-weighted image, T2-weighted image, fluid-attenuated inversion recovery image
Diagnostic Test: Diffusion-weighted MRI — Diffusion-weighted MRI
Diagnostic Test: Arterial spin labeling (ASL) — Cerebral blood flow imaging parameter
Diagnostic Test: Dynamic susceptibility contrast-MRI (DSC-MRI) — Cerebral blood volume and vessel architectural imaging parameters

SUMMARY:
This trial uses multi-parametric magnetic resonance imaging (MRI) to develop and validate imaging risk score to predict radiation necrosis in participants with brain metastasis treated with radiation therapy. Diagnostic procedures, such as multi-parametric magnetic resonance imaging (MRI), may improve the ability to diagnose radiation necrosis early and help establish treatment strategies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop an imaging risk score for recurrence after stereotactic radiosurgery (SRS) in brain metastasis using multiparametric MRI.

II. To validate the imaging risk score in retrospective external validation and prospective internal validation test set.

SECONDARY OBJECTIVE:

I. To predict radiation necrosis using imaging risk score.

OUTLINE:

Participants undergo multi-parametric MRI including 3D pre- and contrast-enhanced T1 weighted image, T2 weighted image, diffusion-weighted image, dynamic susceptibility contrast MRI, and arterial spin labeling image before receiving SRS, and every 3 months after SRS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent stereotactic radiosurgery (SRS, gamma-knife radiosurgery or cyberknife radiosurgery) for brain metastases
2. Patients with lesions eligible for SRS :

   * One to ten newly diagnosed brain metastases
   * Patients without acute neurological symptom
3. Patients with a Karnofsky performance status score of 70 or higher
4. Patients who underwent brain MRI within 1 month of enrollment
5. Patients with measurable enhancing lesions on MRI.
6. Patients who have available reference standard (second-look surgery for recurrence) or available follow up imaging for clinic-radiologic reference standard.
7. A longest diameter > 1.5 cm for tumor habitat analysis.

Exclusion criteria:

1. Patients who have undergone prior brain surgery, SRS, or whole-brain radiation therapy.
2. Patients who are diagnosed with leukemia, lymphoma, germ-cell tumor, small-cell lung cancer, leptomeningeal disease, or unknown primary tumor.
3. Patients with age < 18 years.
4. Patients without baseline MRI.
5. Patients with nonmeasurable enhancing lesions on MRI : all other lesions, including lesions with longest dimension < 10 mm, lesions with borders that cannot be reproducibly measured, dural metastases, bony skull metastases, and leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of tertiary medical center
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Time to progression | up to 24 months
  The time from the date of SRS for brain metastasis until the date of progression.

SECONDARY OUTCOMES:
Response rate | up to 24 months
  The response is determined by response assessment in neuro-oncology brain metastases (RANO-BM) criteria. Clinical and radiologic assessments per lesion and person are carried out at every MRI follow-up using the MRI before SRS as the baseline.
Occurence rate of radiation necrosis | 12 months
  The rate of occurrence of radiation necrosis per lesion is determined through a combination of imaging findings and clinical evaluation by a multidisciplinary team.
Imaging risk score for recurrence | Baseline imaging before SRS, and follow up imaging every 3 months after SRS, up to 24 months
  To calculate the imaging risk score, three parameters are added together, namely the "solid component score," the "less enhancing component score," and the "blood flow score," using contrast-enhanced T1-weighted image(T1WI), T2-weighted image (T2WI), diffusion-weighted imaging (DWI), and ASL.
  The solid component risk score is assigned 0, 1, or 2 points, depending on whether the hypointense lesion on T2WI matches the enhancement in CE-T1WI.
  The less-enhancing component risk score evaluates the degree of enhancement of the lesion to the dura. It assigns 0, 1, or 2 points depending on whether it is brighter, similar, or less enhanced.
  The blood flow risk score assigns 0, 1, or 2 points based on the degree of blood flow of the lesion in ASL.
Tumor habitat analysis | Baseline imaging before SRS, and follow up imaging every 3 months after SRS, up to 24 months
  Automated process of tumor habitat analysis will include followings.
  A. Methods: preprocessing includes registration, deep learning segmentation, and normalization of contrast-enhanced T1-weighted (CE-T1) and T2-weighted images. K-means clustering is applied to CE-T1-weighted and T2-weighted images to construct structural MRI habitats and to apparent diffusion coefficient (ADC) and cerebral blood volume (CBV) images to construct physiologic habitats.
  B. Structural MRI habitats: enhancing tissue habitat, solid low-enhancing habitat, and nonviable tissue habitat
  C. Physiologic MRI habitats: hypervascular cellular habitat, hypovascular cellular habitat, and nonviable tissue habitat..
  D. Quantitative measurement of each habitat will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Le Rhun E, Guckenberger M, Smits M, Dummer R, Bachelot T, Sahm F, Galldiks N, de Azambuja E, Berghoff AS, Metellus P, Peters S, Hong YK, Winkler F, Schadendorf D, van den Bent M, Seoane J, Stahel R, Minniti G, Wesseling P, Weller M, Preusser M; EANO Executive Board and ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. EANO-ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up of patients with brain metastasis from solid tumours. Ann Oncol. 2021 Nov;32(11):1332-1347. doi: 10.1016/j.annonc.2021.07.016. Epub 2021 Aug 6. No abstract available. PMID 34364998
- [Background] Chao ST, Ahluwalia MS, Barnett GH, Stevens GH, Murphy ES, Stockham AL, Shiue K, Suh JH. Challenges with the diagnosis and treatment of cerebral radiation necrosis. Int J Radiat Oncol Biol Phys. 2013 Nov 1;87(3):449-57. doi: 10.1016/j.ijrobp.2013.05.015. Epub 2013 Jun 19. PMID 23790775
- [Background] Jhaveri J, Chowdhary M, Zhang X, Press RH, Switchenko JM, Ferris MJ, Morgan TM, Roper J, Dhabaan A, Elder E, Eaton BR, Olson JJ, Curran WJ, Shu HG, Crocker IR, Patel KR. Does size matter? Investigating the optimal planning target volume margin for postoperative stereotactic radiosurgery to resected brain metastases. J Neurosurg. 2019 Mar 1;130(3):797-803. doi: 10.3171/2017.9.JNS171735. Epub 2018 Apr 20. PMID 29676690
- [Background] Kirkpatrick JP, Wang Z, Sampson JH, McSherry F, Herndon JE 2nd, Allen KJ, Duffy E, Hoang JK, Chang Z, Yoo DS, Kelsey CR, Yin FF. Defining the optimal planning target volume in image-guided stereotactic radiosurgery of brain metastases: results of a randomized trial. Int J Radiat Oncol Biol Phys. 2015 Jan 1;91(1):100-8. doi: 10.1016/j.ijrobp.2014.09.004. Epub 2014 Oct 21. PMID 25442342
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Stockham AL, Tievsky AL, Koyfman SA, Reddy CA, Suh JH, Vogelbaum MA, Barnett GH, Chao ST. Conventional MRI does not reliably distinguish radiation necrosis from tumor recurrence after stereotactic radiosurgery. J Neurooncol. 2012 Aug;109(1):149-58. doi: 10.1007/s11060-012-0881-9. Epub 2012 May 26. PMID 22638727
- [Background] Tsao MN, Rades D, Wirth A, Lo SS, Danielson BL, Gaspar LE, Sperduto PW, Vogelbaum MA, Radawski JD, Wang JZ, Gillin MT, Mohideen N, Hahn CA, Chang EL. Radiotherapeutic and surgical management for newly diagnosed brain metastasis(es): An American Society for Radiation Oncology evidence-based guideline. Pract Radiat Oncol. 2012 Jul-Sep;2(3):210-225. doi: 10.1016/j.prro.2011.12.004. Epub 2012 Jan 30. PMID 25925626
- [Background] Lee DH, Park JE, Kim N, Park SY, Kim YH, Cho YH, Kim HS. Tumor habitat analysis by magnetic resonance imaging distinguishes tumor progression from radiation necrosis in brain metastases after stereotactic radiosurgery. Eur Radiol. 2022 Jan;32(1):497-507. doi: 10.1007/s00330-021-08204-1. Epub 2021 Aug 6. PMID 34357451
- [Background] Park JE, Kim HS, Kim N, Park SY, Kim YH, Kim JH. Spatiotemporal Heterogeneity in Multiparametric Physiologic MRI Is Associated with Patient Outcomes in IDH-Wildtype Glioblastoma. Clin Cancer Res. 2021 Jan 1;27(1):237-245. doi: 10.1158/1078-0432.CCR-20-2156. Epub 2020 Oct 7. PMID 33028594
- [Background] Sneed PK, Mendez J, Vemer-van den Hoek JG, Seymour ZA, Ma L, Molinaro AM, Fogh SE, Nakamura JL, McDermott MW. Adverse radiation effect after stereotactic radiosurgery for brain metastases: incidence, time course, and risk factors. J Neurosurg. 2015 Aug;123(2):373-86. doi: 10.3171/2014.10.JNS141610. Epub 2015 May 15. PMID 25978710
- [Derived] Roh YH, Park JE, Park SY, Cho YH, Kim YH, Song SW, Yoon S, Kim HS. Assessment of imaging risks for recurrence after stereotactic radiosurgery for brain metastases (IRRaS-BM). BMC Cancer. 2024 Jul 18;24(1):866. doi: 10.1186/s12885-024-12636-5. PMID 39026289